CLINICAL TRIAL: NCT01166789
Title: Lubiprostone Effects on Visceral Pain Sensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, William Whitehead, PhD, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-004L
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; pain threshold; constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Active Comparator): Lubiprostone 48ug taken daily for 14 days.
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): 2 capsules containing a substance with no active ingredient taken daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 48ug daily taken as 24ug capsules twice per day, in morning and evening.
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — 2 capsules daily, taken in morning and evening
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine how Lubiprostone, a medication used to treat irritable bowel syndrome with constipation predominant symptoms (IBS-C), works to reduce clinical pain. Lubiprostone acts in the small intestine to cause an increase in the secretion of chloride, water and sodium. The increased fluid causes food residue to move through the bowel more quickly and makes the stools softer. First, we want to test the idea that Lubiprostone works by making a person less sensitive to pain. Second, we want to confirm that Lubiprostone decreases the time it takes fecal matter to travel through your GI tract, referred to as transit time.

DETAILED DESCRIPTION:
Subjects will be enrolled in an 8-week study requiring a total of 7 visits to the UNC Center for Clinical and Translational Research. The protocol is divided into 4 two-week periods: (1) Two-week baseline diary symptom monitoring, followed by a barostat test of pain sensitivity. (2) Two-week treatment with either Lubiprostone or placebo, with daily symptom diary recording and barostat test of pain sensitivity at the end. In addition, patients will be tested for whole gut transit time by the radio-opaque marker (Sitzmark) technique in the second week. (3) Two-week washout period, during which patients will continue the symptom diary. (4) Two-week crossover to Lubiprostone or placebo, identical to the second two-week period.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of IBS-C
* meeting Rome III diagnostic criteria for IBS-C
* age 18 or older

Exclusion Criteria:

* use of laxatives or prokinetics within two weeks prior to the study or during the study
* use of IBS-specific compounds, opiates, anticholinergics, or any drug likely to cause constipation as a side-effect
* use of analgesics for 48 hours prior to the study
* hypothyroid condition
* history of bowel resection except appendectomy or cholecystectomy
* psychotic disorder, major depression, substance abuse (other than tobacco), or other psychiatric condition likely to interfere with the conduct of the study. Subjects treated for depression more than 2 years ago or for situational circumstances may be eligible for the study at the investigator's discretion
* renal disease
* inflammatory or ischemic disease of the rectum
* known to be an unreliable subject
* Because this study involves exposure to radiation, subjects who are pregnant or planning to become pregnant, employees currently working with radiation, and subjects who have participated in research involving radiation within the past year will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pain threshold | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Clinical and Translational Research Center, Chapel Hill, North Carolina, United States